CLINICAL TRIAL: NCT01290978
Title: Prospective, Randomized Comparison of Two Presurgical Skin Antiseptic Preparations and Resultant Surgical Incise Drape Adhesion to Skin
Brief Title: Compare Effect of Surgical Antiseptic Preparations on Incise Drape Adhesion to Skin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: Cyberderm Inc. (Industry); 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 05-011219
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — DuraPrep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ChloraPrep (Active Comparator): Applied ChloraPrep on the application site per manufacturer's instruction
  Interventions: Drug: ChloraPrep
- DuraPrep (Active Comparator): Apply DuraPrep to the application site per manufacturer's instruction
  Interventions: Drug: DuraPrep

INTERVENTIONS:
Drug: ChloraPrep — The application sites (subjects' backs) will be prepped with ChloraPrep according to manufacturer's instruction. Samples of 3 surgical incise drapes will be applied to the prepped sites according to randomization schedule
  Other Names: ChloraPrep® with Tint (Scrub Teal®)
  Arms: ChloraPrep
Drug: DuraPrep — The application sites (subjects' backs) will be prepped with DuraPrep according to manufacturer's instruction. Samples of 3 surgical incise drapes will be applied to the prepped sites according to randomization schedule
  Other Names: 3M™ DuraPrep™ Surgical Solution
  Arms: DuraPrep

SUMMARY:
The purpose of this study is to find out if presurgical antiseptic preparations affect how well surgical drapes adhere to skin.

DETAILED DESCRIPTION:
Adhesive incise drapes are often used to provide a physical sterile barrier between the surrounding skin and the open wound at the beginning of a surgery. This study sought to determine the effect of presurgical skin antiseptic preparation on the adhesion of various incise drapes to the skin.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign the Research Consent form
* Healthy male or female subjects ages between 18 - 65
* Subject has agreed to be and appears to be compliant with requirements of the study
* Subject has a back (the product application site) of sufficient size, free of blemishes to comfortably fit 18 strips of 1/2" x 3" drape samples
* Subject is willing to have the back clipped or shaved if it has excessive hair

Exclusion Criteria:

* Sensitivity/allergy to adhesive products (e.g. medical tapes)
* Sensitivity to the antimicrobial agent iodine, povidone iodine (PVPI), isopropyl alcohol (IPA), or chlorhexidine gluconate (CHG)
* Allergy to seafood
* History of psoriasis dermatitis, or any skin condition that might be exacerbated by the action of removing adhesive materials
* Active dermatitis (rash), sunburn, blemishes, broken skin, cuts, and/or infection on the subject's back
* History of diabetes
* Subject is currently pregnant or thinks she may be pregnant or is nursing
* Subject is receiving steroid-based anti-inflammatory or immunosuppressant drug therapy
* Subject is taking antihistamine medication
* Subject has been using moisturizers or other skin contact materials on the test sites for 24 hours prior to the start of the study
* Subject has a back problem that prohibits him or her from lying face downward for approximately 2 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Grove, PhD, Principal Investigator — Cyberderm Inc.
Locations (1):
- cyberDERM Clinical Studies, Broomall, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted between 22 Feb and 5 March 2010. Twenty-four male or female healthy volunteers between ages of 18 and 65 were screened for this study in order to ensure that at least 20 volunteers were enrolled. Volunteers were recruited from a pool of suburban men/women who met the exclusion/inclusion criteria.
Pre-assignment Details: Volunteers who met the exclusion/inclusion criteria were required to undergo a 1-day washout period where they were not allowed to use any moisturizing products or other skin contact materials on their backs. Two subjects were screen failures.
Groups:
- ChloraPrep, DuraPrep: Subject's back was visually divide into 2. Applied each prep per manufacturer's instruction on either right or left of back according to randomization schedule
Period: Overall Study
Arm/Group | ChloraPrep, DuraPrep
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A sample size of 18 subjects and 18 drape samples per subject was determined to provide 80% power to detect a difference of 20% for the drape by prep comparison. A minimum of 20 subjects was used to account for the uncertainty in variability.
Groups:
- ChloraPrep , DuraPrep: Subject's back was applied with 2 skin preps (ChloraPrep and DuraPrep), one on each side of subject's back per randomization schedule.
Arm/Group | ChloraPrep , DuraPrep
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: participants] | 40.4 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Eleven males and 11 females were enrolled into the study
  Participants
    Female | 11
    Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Drape Adhesion
Description: The peel force to remove the sample
Time Frame: 30 minutes
Population: Data analysis per protocol
Measure: Mean (95% Confidence Interval); unit: grams-force
Groups:
- ChloraPrep; DuraPrep: Subject's back was applied with 2 skin preps (ChloraPrep and DuraPrep), one on each side of subject's back per randomization schedule.
Arm/Group | ChloraPrep | DuraPrep
Number analyzed (Participants) | 22 | 22
grams-force | 78.6 [68.0 to 89.2] | 181.3 [165.8 to 196.8]

2. Secondary Outcome: Skin Assessment on Ioban, ActiGard, Steri-Drape 2 Application Sites Respectively
Description: Visual assessment on skin after samples were removed. scale: 0 (no skin reaction), 4 (severe skin reaction)
Time Frame: 30 minutes
Population: The number of participants was determined to provide 80% power to detect a difference of 20% for the drape by prep comparisons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ChloraPrep | DuraPrep
Number analyzed (Participants) | 22 | 22
units on a scale
  Skin assessment on Ioban application site | 0.67 (0.52) | 0.98 (0.62)
  Skin assessment on ActiGard application site | 0.31 (0.44) | 0.90 (0.65)
  Skin assessment on Steri-Drape 2 application site | 0.30 (0.43) | 0.95 (0.58)

ADVERSE EVENTS:
Arm/Group | ChloraPrep, DuraPrep
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

LIMITATIONS AND CAVEATS:
All 22 subjects enrolled completed the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction for PI to publish trial results without review and approval by sponsor